CLINICAL TRIAL: NCT06041022
Title: A Non-invasive Model to Predict Antiviral Therapy in Patients With Gray Zone of Chronic Hepatitis B: a Multi-center, Retrospective Study
Brief Title: A Non-invasive Model to Predict Antiviral Therapy in Gray Zone of Chronic Hepatitis B
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Linyi People's Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Sir Run Run Shaw Hospital (Other); First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: KYLL-202301-030
Record Dates: First submitted 2023-09-03; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Hepatitis B, Chronic
Keywords: Antiviral therapy; Liver biopsy; Gray zone; Model; Chronic hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Exposure factors — Including demographical data, laboratory features and liver histological indicators.

SUMMARY:
Establishment and validation of the non-invasive model to predict antiviral therapy in the gray zone of chronic hepatitis B

DETAILED DESCRIPTION:
Chronic hepatitis B virus (HBV) infection continues to be a major public health problem worldwide today. According to statistics, the prevalence of chronic HBV infection assessed globally in 2016 was 3.5%, or 257 million people with chronic infection. In China, it is estimated that about 70 million people are chronically infected with HBV in 2019, including about 20-30 million people with chronic hepatitis B (CHB). CHB is a major risk factor for cirrhosis, and hepatocellular carcinoma (HCC). 12-20% of patients with chronic hepatitis B will develop cirrhosis, and of these, around 20% will further develop decompensated cirrhosis and 6-15% will develop HCC, with hepatitis B accounting for approximately 50% of HCC cases worldwide. Therefore, strongly and exact management of chronic hepatitis B is extremely important for the control of HBV progression. Current domestic and international clinical guidelines generally divide the natural history of chronic hepatitis B into four immune phases based on HBV DNA levels, liver injury, and HBeAg status: immune active, immune tolerant, inactive HBsAg carriers, and reactive stage. The guidelines of American Association for the Study of Liver Diseases (AASLD) recommend the use of antiviral therapy for patients in the immune active and reactive phases, and also provide a detailed follow-up plan for patients in other phases. However, a significant number of patients with chronic hepatitis B cannot be classified in any of these four phases, who falls into a gray area with uncertainty of formal management. According to the 2018 AASLD Hepatitis B Guidelines criteria for antiviral therapy, patients in the gray zone still do not have clarity on the need for antiviral therapy based only on clinical indicators. A recent study showed that nearly 40% of patients with chronic hepatitis B were in the indeterminate stage. At long-term follow-up assessment, half of these patients were still in the indeterminate phase and one-fifth had transitioned to the immune active phase. Patients in the indeterminate phase were 14 times more likely to develop HCC than those with inactive hepatitis B. Therefore, the management of antiviral therapy in patients with CHB in the "gray zone" is crucial and should be demonstrated. The aim of the investigators is to investigate the clinical characteristics of patients with uncertain treatment in the "gray zone" of CHB and to develop a non-invasive predictive model for the indication of antiviral therapy. This will provide guidance for the clinical management of patients in the "gray zone" of CHB, thereby reducing the incidence of cirrhosis and liver cancer and improving their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* HBeAg positive, normal serum alanine aminotransferase(ALT) level，HBVDNA≤10^6 IU/ml
* HBeAg positive, elevated serum ALT, HBVDNA≤2*10^4 IU/ml
* HBeAg negative, elevated serum ALT, HBVDNA≤2*10^3 IU/ml
* HBeAg negative, normal serum ALT, HBVDNA≥2*10^3 IU/ml

Normal upper limit of ALT is 35 U/L for male and 25 U/L for female.

Exclusion Criteria:

* Concurrent with other liver diseases such as autoimmune hepatitis, Hepatitis C virus infectious, liver cirrhosis, HCC, or unexplained liver function abnormalities
* Patients with incomplete clinical data

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The minimum sample size required for the study was calculated to be 417, and it was estimated that almost 1000 patients with chronic hepatitis B underwent hepatic puncture biopsy in the seven hospitals from 2010 to 2022, and all patients will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with the antiviral therapy as assessed by AASLD guideline | From Jan 1st,2010 to Aug 31,2023
  The criteria of antiviral therapy:
  1. Immune-active CHB: an elevation of ALT≥2 the upper limit of normal (ULN)plus elevated HBV DNA above 2,000 IU/mL (HBeAg negative) or above 20,000 IU/mL (HBeAg positive).
  2. Immune-active CHB and cirrhosis if HBV DNA is >2,000 IU/mL.
  3. Immune-active CHB with ALT < 2 the ULN and HBV DNA below thresholds (less than 2,000 IU/mL if HBeAg negative or less than 20,000 IU/mL if HBeAg positive) are as follows: 1) Age: older age (>40 years). 2) Family history of cirrhosis or HCC. 3) Previous treatment history. 4) Presence of extrahepatic manifestations. 5) Presence of cirrhosis.
  4. Immune tolerance CHB with the moderate-to-severe necroinflammation or fibrosis on a liver biopsy specimen.
Number of participants with significant liver histology as assessed by Metavia scoring system | From Jan 1st,2010 to Aug 31,2023
  Significant liver histology showing significant hepatic inflammation ≥G2 and/or fibrosis ≥S2 as assessed by Metavir scoring system
  The fibrosis score is used to describe the amount of inflammation (the intensity of inflammation/breakdown of tissue) in the liver:
  F0: No fibrosis F1: Portal fibrosis without septa F2: Portal fibrosis with few septa F3: Numerous septa without cirrhosis F4: Cirrhosis
  The activity score is a prediction about how rapidly the degree of fibrosis is progressing:
  G0: No activity G1: Mild activity G2: Moderate activity G3: Severe activity

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chen Fan, MD,PhD, Study Chair — Qilu Hospital of Shandong University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schweitzer A, Horn J, Mikolajczyk RT, Krause G, Ott JJ. Estimations of worldwide prevalence of chronic hepatitis B virus infection: a systematic review of data published between 1965 and 2013. Lancet. 2015 Oct 17;386(10003):1546-55. doi: 10.1016/S0140-6736(15)61412-X. Epub 2015 Jul 28. PMID 26231459
- [Background] Wang G, Duan Z. Guidelines for Prevention and Treatment of Chronic Hepatitis B. J Clin Transl Hepatol. 2021 Oct 28;9(5):769-791. doi: 10.14218/JCTH.2021.00209. Epub 2021 Sep 28. PMID 34722192
- [Background] Huang DQ, Lim SG. Hepatitis B: Who to treat? A critical review of international guidelines. Liver Int. 2020 Feb;40 Suppl 1:5-14. doi: 10.1111/liv.14365. PMID 32077616
- [Background] Terrault NA, Lok ASF, McMahon BJ, Chang KM, Hwang JP, Jonas MM, Brown RS Jr, Bzowej NH, Wong JB. Update on prevention, diagnosis, and treatment of chronic hepatitis B: AASLD 2018 hepatitis B guidance. Hepatology. 2018 Apr;67(4):1560-1599. doi: 10.1002/hep.29800. No abstract available. PMID 29405329
- [Derived] Ma HY, Yang XY, Tian YX, Li XD, He YL, Yang Q, Zheng MH, Zheng YB, Yu Y, Xu LY, Wang QN, Zhang T, Shi Y, Fan YC. Performance of the AASLD, EASL, and APASL Clinical Practice Guidelines in"grey zone"stages of Chinese patients with chronic hepatitis B. Hepatol Int. 2025 Aug;19(4):796-808. doi: 10.1007/s12072-025-10833-3. Epub 2025 May 14. PMID 40360826
- [Derived] Yang XY, Li XD, Wu BY, Yang Q, Zheng YB, Zheng MH, Wu YP, Ma HY, Zuo J, Jia RX, Yu Y, Xu LY, Tian YX, An Q, Zhang T, He YL, Shi Y, Fan YC. A Model to Identify Gray Zone Patients With Chronic Hepatitis B Requiring Antiviral Therapy: A Multicenter Retrospective Study. J Infect Dis. 2025 Aug 14;232(2):485-498. doi: 10.1093/infdis/jiaf070. PMID 39960318